CLINICAL TRIAL: NCT00990197
Title: The Safety of Transdermal Nicotine Immediately Following an Acute Coronary Syndrome: The STADIA Pilot Study
Brief Title: The Safety of Transdermal Nicotine Immediately Following an Acute Coronary Syndrome
Acronym: STADIA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with enrollment.
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Canadian Tobacco Control Research Initiative (Other)
Responsible Party: Mark J. Eisenberg, MD MPH, Jewish General Hospital/McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-023; 016026
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Smoking Cessation
Keywords: Pilot study; Randomized clinical trial; Smoking cessation; Acute coronary syndrome; Transdermal nicotine patch
MeSH Terms: conditions — Smoking Cessation; Acute Coronary Syndrome | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day 1 (Active Comparator): Patients randomized to wearing the patch on day 1 will apply a patch on the morning of their treatment day and keep it on for 24 hours. These patients will not wear a patch on day 2.
  Interventions: Drug: Transdermal nicotine patch
- Day 2 (Active Comparator): Patients randomized to wearing the patch on day 2 will apply a patch on the morning of their treatment day and keep it on for 24 hours. These patients will not wear a patch on day 1.
  Interventions: Drug: Transdermal nicotine patch

INTERVENTIONS:
Drug: Transdermal nicotine patch — Subjects will apply the nicotine patch on the morning of their treatment day and will keep it on for 24 hours.
  Other Names: Nicoderm CQ, Biovail Pharmaceuticals

SUMMARY:
Continuing to smoke after having a heart attack greatly increases the risk of death and cardiac illness. The nicotine patch is a commonly used pharmacotherapy for smoking cessation and has great potential to help heart attack patients quit smoking. However, due to safety concerns, physicians are often hesitant to prescribe the nicotine patch to patients who have just suffered a heart attack. The STADIA pilot study will assess the feasibility of a large-scale clinical trial investigating safety and efficacy outcomes associated with the nicotine patch immediately following a heart attack. Eligible subjects will be randomized within 48 hours of suffering a heart attack to wear a transdermal nicotine patch on either day 1 or day 2 of the study period. The nicotine patch will deliver nicotine to the patient over the period of 24 hours. Patients will be advised to discuss smoking cessation strategies with their treating physician and subsequent care will be left to the discretion of this physician. The duration of ischemia (loss of blood flow in the heart), patient adherence, incidence of arrhythmia (disorder of the heart rate or rhythm), heart rate, and blood pressure within the two groups will be used to evaluate the safety of transdermal nicotine use immediately after a heart attack.

DETAILED DESCRIPTION:
Objective

The STADIA Pilot Study will be used to evaluate the feasibility of conducting a three-year multi-centre trial investigating the long-term safety and efficacy outcomes associated with transdermal nicotine use immediately following an acute coronary syndrome (ACS).

Rationale

Patients who initially survive an ACS are at high risk of recurrent cardiac events or cardiovascular death. Within the first 6 months alone, 12% of patients will die or suffer another ACS, while another 23% will require revascularization for angina. Patients who are able to quit smoking reduce their chances of suffering a recurrent ACS or cardiovascular death within the next year by ≥ 50%. After surviving an ACS, most patients are highly motivated to stop smoking. However, as nicotine is an extremely addictive psychoactive drug, up to 60% of patients who attempt to quit relapse. Hospitalization following an ACS provides an opportunity for smokers to quit, as smoking while in hospital is prohibited. However, abstinence while hospitalized also precipitates intense nicotine withdrawal symptoms, which are largely responsible for the high rates of smoking relapse. Nicotine replacement therapy (NRT) can ameliorate many of these symptoms and increase the chances that smokers continue to abstain from tobacco use after discharge. Of the available NRTs, transdermal nicotine is associated with the least severe cardiovascular effects, as it delivers nicotine more gradually (with lower peak values) than nicotine gum or inhalers. Although transdermal nicotine more than doubles long-term smoking cessation rates when compared with placebo, it is rarely prescribed by physicians in the weeks immediately following an ACS because the possible cardiovascular effects of nicotine after an ACS have yet to be systematically evaluated.

Methods

A total of 30 patients will be randomized within 48-hours of suffering an ACS from the Jewish General Hospital (Montreal, QC) and collaborating centres. Prior to randomization, all patients will receive standardized smoking cessation counselling. Subjects who satisfy the inclusion and exclusion criteria for the trial will be randomized within 48 hours of suffering an ACS to wear a transdermal nicotine patch on either day 1 or day 2 of the study period. Subjects will apply a patch the morning of their treatment day and keep it on for 24 hours. Patients will be advised to discuss smoking cessation strategies with their treating physician and subsequent care will be left to the discretion of this physician. Twenty-four hour Holter monitoring will be used to measure heart rate, incidence of arrhythmia, and the duration of ischemic events at day 1 and day 2 of the study period. Systolic and diastolic blood pressure will be assessed via 24-hour Ambulatory blood pressure monitoring (ABPM). ABPM will be used on day 1 and day 2 of the study period. On day 1 the study nurse will record the severity of nicotine withdrawal symptoms, side effects, any smoking relapses and if so, how many cigarettes were smoked, and any medications they are currently taking. On day 7 and 14 patients will be contacted by telephone to determine the severity of nicotine withdrawal symptoms, any smoking relapses and if so, how many cigarettes were smoked and any medications they are currently taking. Cardiovascular events will be assessed by patient monitoring and by a study nurse. Nicotine withdrawal symptoms according to the Hughes-Hatsukami symptom scale and common nicotine patch side effects, severity-rated on a five-point scale, will be determined through study nurse inquiries on days 1, 7, and 14 (6). Carbon monoxide monitors will be used to measure levels of expired CO at baseline. Participants whose levels of expired CO exceed 10 ppm will be classified as smokers.

Significance

If shown to be safe and effective, transdermal nicotine will have a major impact on the secondary prevention of recurrent cardiac events on the 20,000 Canadian smokers who suffer an ACS each year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Current smoker, ≥ 10 cigarettes per day, on average, for the past year
* Suffered an enzyme-positive ACS (Troponin T, Troponin I, or CK-MD) and planned hospitalization of ≥ 48 hours
* Motivated to quit smoking

Exclusion Criteria:

* Current use of any medical therapy for smoking cessation
* History of alcohol or controlled substance abuse
* History of severe dermatitis
* Current diagnosis of unstable psychiatric illness requiring medication
* Suffered an ACS as a complication of a hospitalization for a different condition (i.e. postoperatively)
* Pregnancy or lactation
* Likely to be unavailable for follow-up
* Unable to read and understand English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The total duration of ischemic episodes | Day 1 and Day 2

SECONDARY OUTCOMES:
Patient adherence to study protocol | Day 1, Day 7, Day 14
Incidence of arrhythmia | Day 1 and Day 2
Heart rate | Day 1 and Day 2
Systolic and diastolic blood pressure | Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Eisenberg, MD MPH, Principal Investigator — Jewish General Hospital/McGill University
Locations (1):
- SMDB Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Sauer WH, Berlin JA, Strom BL, Miles C, Carson JL, Kimmel SE. Cigarette yield and the risk of myocardial infarction in smokers. Arch Intern Med. 2002 Feb 11;162(3):300-6. doi: 10.1001/archinte.162.3.300. PMID 11822922
- [Background] Cardiovascular Disease Surveillance. Laboratory Centre for Disease Control, Statistics Canada 2002, Candian Institutes for Health Information (CIHI), 2002.
- [Background] Nicotine replacement therapy for patients with coronary artery disease. Working Group for the Study of Transdermal Nicotine in Patients with Coronary artery disease. Arch Intern Med. 1994 May 9;154(9):989-95. PMID 8179456
- [Background] Frid D, Ockene IS, Ockene JK, Merriam P, Goldberg R, Kristeller J, Barrett S. Severity of angiographically proven coronary artery disease predicts smoking cessation. Am J Prev Med. 1991 May-Jun;7(3):131-5. PMID 1931139
- [Background] Brummett BH, Babyak MA, Mark DC, Williams RB, Siegler IC, Clapp-Channing N, Barefoot JC. Predictors of smoking cessation in patients with a diagnosis of coronary artery disease. J Cardiopulm Rehabil. 2002 May-Jun;22(3):143-7. doi: 10.1097/00008483-200205000-00003. PMID 12042680
- [Background] Hughes JR. Tobacco withdrawal in self-quitters. J Consult Clin Psychol. 1992 Oct;60(5):689-97. doi: 10.1037//0022-006x.60.5.689. PMID 1401384
- [Background] Stapleton J. Cigarette smoking prevalence, cessation and relapse. Stat Methods Med Res. 1998 Jun;7(2):187-203. doi: 10.1177/096228029800700206. PMID 9654641
- [Background] Rigotti NA, Arnsten JH, McKool KM, Wood-Reid KM, Pasternak RC, Singer DE. Smoking by patients in a smoke-free hospital: prevalence, predictors, and implications. Prev Med. 2000 Aug;31(2 Pt 1):159-66. doi: 10.1006/pmed.2000.0695. PMID 10938217
- [Background] Jorenby DE, Hatsukami DK, Smith SS, Fiore MC, Allen S, Jensen J, Baker TB. Characterization of tobacco withdrawal symptoms: transdermal nicotine reduces hunger and weight gain. Psychopharmacology (Berl). 1996 Nov;128(2):130-8. doi: 10.1007/s002130050118. PMID 8956374
- [Background] Benowitz NL, Fitzgerald GA, Wilson M, Zhang Q. Nicotine effects on eicosanoid formation and hemostatic function: comparison of transdermal nicotine and cigarette smoking. J Am Coll Cardiol. 1993 Oct;22(4):1159-67. doi: 10.1016/0735-1097(93)90431-y. PMID 7691912
- [Background] Mulligan SC, Masterson JG, Devane JG, Kelly JG. Clinical and pharmacokinetic properties of a transdermal nicotine patch. Clin Pharmacol Ther. 1990 Mar;47(3):331-7. doi: 10.1038/clpt.1990.36. PMID 2311334
- [Background] Gourlay S. The pros and cons of transdermal nicotine therapy. Med J Aust. 1994 Feb 7;160(3):152-9. PMID 8295585
- [Background] Benowitz NL. Drug therapy. Pharmacologic aspects of cigarette smoking and nicotine addiction. N Engl J Med. 1988 Nov 17;319(20):1318-30. doi: 10.1056/NEJM198811173192005. No abstract available. PMID 3054551
- [Background] Kaijser L, Berglund B. Effect of nicotine on coronary blood-flow in man. Clin Physiol. 1985 Dec;5(6):541-52. doi: 10.1111/j.1475-097x.1985.tb00767.x. PMID 4092414
- [Background] Transdermal nicotine for smoking cessation. Six-month results from two multicenter controlled clinical trials. Transdermal Nicotine Study Group. JAMA. 1991 Dec 11;266(22):3133-8. PMID 1956099
- [Background] Pickering TG, Schwartz JE, James GD. Ambulatory blood pressure monitoring for evaluating the relationships between lifestyle, hypertension and cardiovascular risk. Clin Exp Pharmacol Physiol. 1995 Mar;22(3):226-31. doi: 10.1111/j.1440-1681.1995.tb01986.x. PMID 7554420
- [Background] Palatini P, Pessina AC, Graniero GR, Canali C, Mormino P, Dorigatti F, Accurso V, Michieletto M, Ferrarese E, Vriz O, et al. [The relationship between overweight, life style and casual and 24-hour pressures in a population of male subjects with mild hypertension. The results of the HARVEST study]. G Ital Cardiol. 1995 Aug;25(8):977-89. Italian. PMID 7498631
- [Background] Zevin S, Jacob P 3rd, Benowitz NL. Dose-related cardiovascular and endocrine effects of transdermal nicotine. Clin Pharmacol Ther. 1998 Jul;64(1):87-95. doi: 10.1016/S0009-9236(98)90026-1. PMID 9695723
- [Background] Mahmarian JJ, Moye LA, Nasser GA, Nagueh SF, Bloom MF, Benowitz NL, Verani MS, Byrd WG, Pratt CM. Nicotine patch therapy in smoking cessation reduces the extent of exercise-induced myocardial ischemia. J Am Coll Cardiol. 1997 Jul;30(1):125-30. doi: 10.1016/s0735-1097(97)00128-9. PMID 9207632
- [Background] Longo LD. The biological effects of carbon monoxide on the pregnant woman, fetus, and newborn infant. Am J Obstet Gynecol. 1977 Sep 1;129(1):69-103. doi: 10.1016/0002-9378(77)90824-9. No abstract available. PMID 561541
- [Background] Rietbrock N, Kunkel S, Worner W, Eyer P. Oxygen-dissociation kinetics in the blood of smokers and non-smokers: interaction between oxygen and carbon monoxide at the hemoglobin molecule. Naunyn Schmiedebergs Arch Pharmacol. 1992 Jan;345(1):123-8. doi: 10.1007/BF00175479. PMID 1538790
- [Background] Allred EN, Bleecker ER, Chaitman BR, Dahms TE, Gottlieb SO, Hackney JD, Pagano M, Selvester RH, Walden SM, Warren J. Short-term effects of carbon monoxide exposure on the exercise performance of subjects with coronary artery disease. N Engl J Med. 1989 Nov 23;321(21):1426-32. doi: 10.1056/NEJM198911233212102. PMID 2682242
- [Background] Allen SS, Hatsukami D, Gorsline J. Cholesterol changes in smoking cessation using the transdermal nicotine system. Transdermal Nicotine Study Group. Prev Med. 1994 Mar;23(2):190-6. doi: 10.1006/pmed.1994.1026. PMID 8047525
- [Background] Morrow JD, Frei B, Longmire AW, Gaziano JM, Lynch SM, Shyr Y, Strauss WE, Oates JA, Roberts LJ 2nd. Increase in circulating products of lipid peroxidation (F2-isoprostanes) in smokers. Smoking as a cause of oxidative damage. N Engl J Med. 1995 May 4;332(18):1198-203. doi: 10.1056/NEJM199505043321804. PMID 7700313
- [Background] Peters RW, Benowitz NL, Valenti S, Modin G, Fisher ML. Electrophysiologic effects of cigarette smoking in patients with and without chronic beta-blocker therapy. Am J Cardiol. 1987 Nov 1;60(13):1078-82. doi: 10.1016/0002-9149(87)90356-0. PMID 2890291
- [Background] Gillum RF, Ingram DD, Makuc DM. White blood cell count and stroke incidence and death. The NHANES I epidemiologic follow-up study. Am J Epidemiol. 1994 May 1;139(9):894-902. doi: 10.1093/oxfordjournals.aje.a117095. PMID 8166139
- [Background] Grimm RH Jr, Neaton JD, Ludwig W. Prognostic importance of the white blood cell count for coronary, cancer, and all-cause mortality. JAMA. 1985 Oct 11;254(14):1932-7. PMID 4046122
- [Background] Hansen PR. Role of neutrophils in myocardial ischemia and reperfusion. Circulation. 1995 Mar 15;91(6):1872-85. doi: 10.1161/01.cir.91.6.1872. PMID 7882499
- [Background] Barnes PJ. New concepts in chronic obstructive pulmonary disease. Annu Rev Med. 2003;54:113-29. doi: 10.1146/annurev.med.54.101601.152209. Epub 2001 Dec 3. PMID 12359824
- [Background] Zevin S, Benowitz NL. Drug interactions with tobacco smoking. An update. Clin Pharmacokinet. 1999 Jun;36(6):425-38. doi: 10.2165/00003088-199936060-00004. PMID 10427467
- [Background] Dacosta A, Guy JM, Tardy B, Gonthier R, Denis L, Lamaud M, Cerisier A, Verneyre H. Myocardial infarction and nicotine patch: a contributing or causative factor? Eur Heart J. 1993 Dec;14(12):1709-11. doi: 10.1093/eurheartj/14.12.1709. PMID 8131771
- [Background] Warner JG Jr, Little WC. Myocardial infarction in a patient who smoked while wearing a nicotine patch. Ann Intern Med. 1994 Apr 15;120(8):695. doi: 10.7326/0003-4819-120-8-199404150-00023. No abstract available. PMID 8135462
- [Background] Ottervanger JP, Festen JM, de Vries AG, Stricker BH. Acute myocardial infarction while using the nicotine patch. Chest. 1995 Jun;107(6):1765-6. doi: 10.1378/chest.107.6.1765. PMID 7781384
- [Background] Hwang SL WM. Heart attacks reported in patch users still smoking. Wall Street Journal 1992;(June 19):B1.
- [Background] Fredrickson PA, Hurt RD, Lee GM, Wingender L, Croghan IT, Lauger G, Gomez-Dahl L, Offord KP. High dose transdermal nicotine therapy for heavy smokers: safety, tolerability and measurement of nicotine and cotinine levels. Psychopharmacology (Berl). 1995 Dec;122(3):215-22. doi: 10.1007/BF02246542. PMID 8748390
- [Background] Pierce JR Jr. Stroke following application of a nicotine patch. Ann Pharmacother. 1994 Mar;28(3):402. doi: 10.1177/106002809402800320. No abstract available. PMID 8193434
- [Background] Jackson M. Cerebral arterial narrowing with nicotine patch. Lancet. 1993 Jul 24;342(8865):236-7. doi: 10.1016/0140-6736(93)92323-l. No abstract available. PMID 8100951
- [Background] Jorenby DE, Smith SS, Fiore MC, Hurt RD, Offord KP, Croghan IT, Hays JT, Lewis SF, Baker TB. Varying nicotine patch dose and type of smoking cessation counseling. JAMA. 1995 Nov 1;274(17):1347-52. PMID 7563558
- [Background] Arnaot MR. Treating heart disease. Nicotine patches may not be safe. BMJ. 1995 Mar 11;310(6980):663-4. doi: 10.1136/bmj.310.6980.663c. No abstract available. PMID 7703770
- [Background] Treating tobacco dependence: a report of the Surgeon General. Washington, DC: Department of Health and Human Services, 2000.
- [Background] Freedman D PRPR. Statistics. New York: Norton Publishers, 1978.
- [Background] Wilson K, Gibson N, Willan A, Cook D. Effect of smoking cessation on mortality after myocardial infarction: meta-analysis of cohort studies. Arch Intern Med. 2000 Apr 10;160(7):939-44. doi: 10.1001/archinte.160.7.939. PMID 10761958
- [Background] Tang JL, Law M, Wald N. How effective is nicotine replacement therapy in helping people to stop smoking? BMJ. 1994 Jan 1;308(6920):21-6. doi: 10.1136/bmj.308.6920.21. PMID 8179658
- [Background] Fiore MC, Smith SS, Jorenby DE, Baker TB. The effectiveness of the nicotine patch for smoking cessation. A meta-analysis. JAMA. 1994 Jun 22-29;271(24):1940-7. PMID 8201739
- [Background] Silagy C, Mant D, Fowler G, Lodge M. Meta-analysis on efficacy of nicotine replacement therapies in smoking cessation. Lancet. 1994 Jan 15;343(8890):139-42. doi: 10.1016/s0140-6736(94)90933-4. PMID 7904003
- [Background] Fiore MC. US public health service clinical practice guideline: treating tobacco use and dependence. Respir Care. 2000 Oct;45(10):1200-62. PMID 11054899
- [Background] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2001;(3):CD000146. doi: 10.1002/14651858.CD000146. PMID 11686953
- [Background] Hughes JR, Glaser M. Transdermal nicotine for smoking cessation. Health Values 1993; 17(2):25-31.
- [Background] American Medical Association. Drug Evaluations Annual 1994. Chicago: American Medical Association 1993.
- [Background] Palmer KJ, Buckley MM, Faulds D. Transdermal Nicotine. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic efficacy as an aid to smoking cessation. Drugs. 1992 Sep;44(3):498-529. doi: 10.2165/00003495-199244030-00011. PMID 1382940
- [Background] Greenland S, Satterfield MH, Lanes SF. A meta-analysis to assess the incidence of adverse effects associated with the transdermal nicotine patch. Drug Saf. 1998 Apr;18(4):297-308. doi: 10.2165/00002018-199818040-00005. PMID 9565740
- [Background] Joseph AM, Norman SM, Ferry LH, Prochazka AV, Westman EC, Steele BG, Sherman SE, Cleveland M, Antonuccio DO, Hartman N, McGovern PG. The safety of transdermal nicotine as an aid to smoking cessation in patients with cardiac disease. N Engl J Med. 1996 Dec 12;335(24):1792-8. doi: 10.1056/NEJM199612123352402. PMID 8943160
- [Background] Tzivoni D, Keren A, Meyler S, Khoury Z, Lerer T, Brunel P. Cardiovascular safety of transdermal nicotine patches in patients with coronary artery disease who try to quit smoking. Cardiovasc Drugs Ther. 1998 Jul;12(3):239-44. doi: 10.1023/a:1007757530765. PMID 9784902
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Moyer D. Chapter 13: Physical fitness and carbon monoxide. Tobacco Reference Guide 2000;30-34.